CLINICAL TRIAL: NCT03266549
Title: Botulinum Toxin Augmented Surgery Versus Conventional Surgery in the Management of Large Angle Concomitant Horizontal Deviations
Brief Title: Botulinum Toxin Augmented Surgery vs Conventional Surgery in the Management of Large Angle Horizontal Deviations
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Sara Alattar, MD, assistant lecturer, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Botox Horizontal Strabismus
Record Dates: First submitted 2017-08-26; First posted 2017-08-30 (Actual); Last update posted 2021-02-21 (Actual); Status verified 2021-02

CONDITIONS: Large Angle Horizontal Strabismus
Keywords: botulinum toxin; horizontal strabismus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Botulinum toxin augmented surgery group (Experimental): unilateral recess-resect procedure, or bilateral rectus muscle recession plus intraoperative injection of 2.5 to 5 units of botulinum toxin A into the recessed muscle.
  Interventions: Procedure: botulinum toxin augmented surgery
- conventional surgery group (Active Comparator): unilateral recess-resect procedure, bilateral rectus muscle recession, or 3 horizontal rectus muscle surgery according to the type of strabismus and the presence or absence of deep amblyopia.The standard correction tables will be used as a guide for the amount of muscle recession and, or resection
  Interventions: Procedure: conventional surgery

INTERVENTIONS:
Procedure: botulinum toxin augmented surgery — unilateral recess-resect procedure, or bilateral rectus muscle recession plus intraoperative injection of 2.5 to 5 units of botulinum toxin A into the recessed muscle.
  Arms: Botulinum toxin augmented surgery group
Procedure: conventional surgery — unilateral recess-resect procedure, bilateral rectus muscle recession, or 3 horizontal rectus muscle surgery according to the type of strabismus and the presence or absence of deep amblyopia. The standard correction tables will be used as a guide for the amount of muscle recession and, or resection.
  Arms: conventional surgery group

SUMMARY:
Horizontal strabismus includes esotropia and exotropia where there is inward or outward deviation of visual axes of the eyes respectively. The most common initial treatment of horizontal strabismus is either bilateral rectus muscle recessions or unilateral recession resection surgery. For large angle deviations (>50 prism diopters [PD]), surgery on 2 muscles alone may not be adequate with high reoperation rates. Approaches to these patients included large bilateral muscle recessions, supramaximal unilateral recession resection procedure, three or four horizontal muscle surgery, or botulinum toxin augmented surgery.

Botulinum toxin augmentated strabismus surgery was reported in several studies. Owens et al.reported successful botulinum toxin augmentation of monocular recession-resection surgeries in 3 large-angle exotropia patients with successful results in two of the 3 patients. Khan reported 8 patients with > 60 PD esotropia treated with botulinum-augmented surgery. Six of 8 had deviations of 10 PD or less following surgery. Özkan et al used botulinum augmentation in a group of older patients with large angle esotropia of different etiologies, with a success rate of 57%. Lueder et al evaluated the long-term outcomes in patients with infantile esotropia. The results were good, with a 74% success rate. Based on historical comparisons, this technique appears equally as effective as 3- or 4-muscle surgery and more effective than large bilateral medial rectus recessions alone.

Ideally, a prospective randomized study should be performed to more definitively determine the effectiveness of intraoperative botulinum toxin augmentation compared to surgery alone.

DETAILED DESCRIPTION:
Strabismus is defined as inability of the two eyes to align their visual axes to a common object of regard. Horizontal strabismus may be in the form of esotropia or exotropia depending on whether the visual axes and the eyes are converging or diverging respectively.

There are multiple surgical techniques used to treat horizontal strabismus with the main goal being to align the visual axes so that binocular vision may develop. The most common initial treatment is either bilateral rectus muscle recessions or unilateral recession resection surgery. For large angle deviations (>50 prism diopters [PD]), surgery on 2 muscles alone may not be adequate to correct the strabismus with high reoperation rates. Approaches to these patients have included large bilateral muscle recessions, supramaximal unilateral recession resection procedure, three or four horizontal muscle surgery, or botulinum toxin augmented surgery.

Botulinum toxin exerts its effect by interfering with release of acetylcholine at the neuromuscular junction, thus inhibiting muscle contraction. Although the pharmacologic effect of botulinum toxin is temporary, permanent results in patients with strabismus may occur. These effects include a change in the length-tension curves of the muscles and permanent changes in sarcomere density and myosin heavy chain composition.

Botulinum toxin alone has been advocated by McNeer and associates as a primary treatment for infantile esotropia in children with smaller angles of deviation. The advantage of this approach is that incisional surgery is not required. However, it was found that botulinum alone was less effective in establishing binocularity when compared to standard surgery. This is likely because multiple injections are often needed, which prolongs the duration of misalignment. On the other hand, the concomitant use of botulinum toxin and surgery allowed for rapid establishment of alignment. Other advantages of botulinum augmentation are that only 2 muscles are operated upon, thus decreasing anesthesia duration and the risk of surgical complications, and the lateral rectus muscles are preserved for additional surgery, if needed.

Botulinum toxin augmentation of strabismus surgery was reported in several previous studies. Owens et al. reported the successful intraoperative use of botulinum toxin to augment monocular recession-resection surgeries in three large-angle exotropia patients. Two of these patients had orthotropia ±10 PD at their final examinations, while the third patient demonstrated a stable 18 PD exotropia which was cosmetically satisfactory. Khan reported 8 patients with > 60 PD esotropia treated with botulinum-augmented horizontal muscle surgery. Six of 8 had deviations of 10 PD or less following surgery, with an average follow-up of 9 months. Özkan et al. used botulinum augmentation in a group of older patients (age range 5-50 years) with large-angle esotropia of different etiologies, with a success rate of 57% and an average follow-up of 14 months. Minguini et al. compared the results of surgery alone versus surgery plus treatment with botulinum toxin for treatment of 23 patient with large angle strabismus. Lueder et al. evaluated the long-term outcomes in patients with infantile esotropia who had been followed for more than 2 years after treatment. The results were good, with a 74% success rate. This study demonstrated that this procedure is an effective treatment for infants with large-angle infantile esotropia, with stable results over time2. Based on historical comparisons, it appears equally as effective as 3- or 4-muscle surgery and more effective than large bilateral medial rectus recessions alone.

Ideally, a prospective randomized study should be performed to more definitively determine the effectiveness of the addition of intraoperative botulinum toxin compared to surgery alone.

ELIGIBILITY:
Inclusion Criteria:

* Large angle concomitant horizontal strabismus (>50 prism diopters)

Exclusion Criteria:

* Other neurologic, or developmental disorders
* Vertical deviation
* Significant A or V patterns
* Paralytic or restrictive forms of strabismus
* History of eye surgery (strabismus or otherwise)

Min Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2021-02-20 (Estimated); Primary Completion 2021-08-31 (Estimated); Study Completion 2021-11-30 (Estimated)

PRIMARY OUTCOMES:
success rate | Patients will be examined at 1 week after surgery
  Outcomes will be considered successful if the patients had orthotropia ±10 PD

SECONDARY OUTCOMES:
incidence of complications | Patients will be examined at 1 week after surgery
  ptosis vertical deviation under-correction (residual esotropia) overcorrection (consecutive exotropia)
Ocular alignment | 12 months postoperative
  Orthotropia or angle of deviation if present

CONTACTS AND LOCATIONS:
Overall Officials: sara Alattar, Principal Investigator — Assiut University
Locations (1):
- Ophthalmology department, faculty of medicine, Assiut university, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lueder GT, Galli M, Tychsen L, Yildirim C, Pegado V. Long-term results of botulinum toxin-augmented medial rectus recessions for large-angle infantile esotropia. Am J Ophthalmol. 2012 Mar;153(3):560-3. doi: 10.1016/j.ajo.2011.08.019. Epub 2011 Oct 13. PMID 21996305
- [Background] Vroman DT, Hutchinson AK, Saunders RA, Wilson ME. Two-muscle surgery for congenital esotropia: rate of reoperation in patients with small versus large angles of deviation. J AAPOS. 2000 Oct;4(5):267-70. doi: 10.1067/mpa.2000.106960. PMID 11040475
- [Background] Bayramlar H, Karadag R, Yildirim A, Ocal A, Sari U, Dag Y. Medium-term outcomes of three horizontal muscle surgery in large-angle infantile esotropia. J Pediatr Ophthalmol Strabismus. 2014 May-Jun;51(3):160-4. doi: 10.3928/01913913-20140318-02. Epub 2014 Mar 25. PMID 24654800
- [Background] Minkoff OV, Donahue SP. Three-muscle surgery for infantile esotropia in children younger than age 2 years. J Pediatr Ophthalmol Strabismus. 2005 May-Jun;42(3):144-8; qiuz 174-5. doi: 10.3928/01913913-20050501-01. PMID 15977866
- [Background] Khan AO. Two horizontal rectus eye muscle surgery combined with botulinum toxin for the treatment of very large angle esotropia. A pilot study. Binocul Vis Strabismus Q. 2005;20(1):15-20. PMID 15828866
- [Background] Ozkan SB, Topaloglu A, Aydin S. The role of botulinum toxin A in augmentation of the effect of recession and/or resection surgery. J AAPOS. 2006 Apr;10(2):124-7. doi: 10.1016/j.jaapos.2005.11.011. PMID 16678746
- [Background] McNeer KW, Tucker MG, Spencer RF. Botulinum toxin management of essential infantile esotropia in children. Arch Ophthalmol. 1997 Nov;115(11):1411-8. doi: 10.1001/archopht.1997.01100160581010. PMID 9366672
- [Background] Owens PL, Strominger MB, Rubin PA, Veronneau-Troutman S. Large-angle exotropia corrected by intraoperative botulinum toxin A and monocular recession resection surgery. J AAPOS. 1998 Jun;2(3):144-6. doi: 10.1016/s1091-8531(98)90004-0. PMID 10532749
- [Background] Minguini N, de Carvalho KM, Bosso FL, Hirata FE, Kara-Jose N. Surgery with intraoperative botulinum toxin-A injection for the treatment of large-angle horizontal strabismus: a pilot study. Clinics (Sao Paulo). 2012;67(3):279-82. doi: 10.6061/clinics/2012(03)13. No abstract available. PMID 22473411